CLINICAL TRIAL: NCT06719128
Title: An Open-Label, Nonrandomized, Single-Dose, Safety and Pharmacokinetic Study of LY3537982 in Participants With Hepatic Impairment and Healthy Participants
Brief Title: A Study of Olomorasib (LY3537982) in Participants With Hepatic Impairment and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18677; J3M-OX-JZQF (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Insufficiency; Healthy
Keywords: Olomorasib; Hepatic Impairment
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Olomorasib (Mild Hepatic Impairment) (Experimental): Olomorasib administered orally.
  Interventions: Drug: Olomorasib
- Olomorasib (Moderate Hepatic Impairment) (Experimental): Olomorasib administered orally.
  Interventions: Drug: Olomorasib
- Olomorasib (Severe Hepatic Impairment) (Experimental): Olomorasib administered orally.
  Interventions: Drug: Olomorasib
- Olomorasib (Normal Hepatic Function) (Experimental): Olomorasib administered orally.
  Interventions: Drug: Olomorasib

INTERVENTIONS:
Drug: Olomorasib — Administered orally.
  Other Names: LY3537982

SUMMARY:
The main purpose of this study is to assess how olomorasib gets into the blood stream and how long it takes the body to remove it when administered to participants with mild, moderate and severe impaired liver function compared to participants with normal liver function. The safety and tolerability of olomorasib will also be evaluated. The study may last up to 6 weeks for each participant including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential.
* Men or women with a body mass index of 18.0 to 40.0 kilograms per meter squared (kg/m²).
* Able to comply with all study procedures, including the 5- to 6-night stays at the CRU and the follow-up phone call.
* Healthy participants: In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, or clinical laboratory evaluations at screening and/or admission as assessed by the investigator (or designee).
* Participants with hepatic impairment: Diagnosis of cirrhosis due to parenchymal liver disease, which is confirmed and documented by at least one of the following: medical history, physical examination, hepatic ultrasound, computed axial tomography scan, magnetic resonance imaging, and/or liver biopsy.

Exclusion Criteria:

* Females who are lactating or of childbearing potential.
* History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:

  1. Metabolic disease
  2. Gastrointestinal disease
  3. Hematological disease
  4. Neurological disease
  5. History or presence of clinically significant cardiovascular disease.
* Abnormal laboratory values determined to be clinically significant by the Investigator (or designee).
* Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination.
* Participation in any other investigational study drug trial involving administration of any investigational drug in the past 30 days or 5 half-lives, whichever was longer, prior to the first dose administration (Day 1).
* Use or intention to use any prescription or over-the-counter medications within 14 days prior to the first dose administration (Day 1) and through end of trial, unless deemed acceptable by the investigator (or designee) and medical monitor.
* History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the participant at undue risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum observed concentration (Cmax) of Olomorasib | Predose on Day 1 up to 96 hours postdose
  PK: Cmax of Olomorasib
PK: Area under the concentration versus time curve from time zero to infinity (AUC0-inf) of Olomorasib | Predose on Day 1 up to 96 hours postdose
  PK: AUC0-inf of Olomorasib

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Orange County Research Center, Lake Forest, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No